CLINICAL TRIAL: NCT03274362
Title: Evaluating the Effectiveness of Headspace Mindfulness Application Versus Standard Care on the HbA1C and Quality of Life in Patients With Diabetes: A Randomized Control Trial
Brief Title: Headspace Mindfulness App Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BCDiabetes.Ca (Network)
Responsible Party: Principal Investigator, Tom Elliott, Medical Director, BCDiabetes.Ca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCDiabetes
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study will use a parallel study model that consists of a treatment arm (ie. Headspace mindfulness app group) and a control arm (ie. standard care where patients receive a list of resources on mindfulness and health).
Masking Description: The study is a prospective, randomized, non-blinded comparative group clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Headspace Application Treatment Group (Experimental): Participants in the treatment group will be given a free 3-month access code to Headspace. The app contains a series of sessions that guide the user through mindfulness training.
  Interventions: Behavioral: Headspace Mindfulness App
- Standard Care Control Group (No Intervention): Participants in the control group will be provided a list of resources that provides guidance on mindfulness and general health.

INTERVENTIONS:
Behavioral: Headspace Mindfulness App — Participants will be given instructions on how to download Headspace on an electronic device and will be provided a free 3-month access code. The app contains a series of ten step-wise 10-minute video sessions that guide the user through mindfulness training. Upon completion of these sessions, additional content will be accessible, including sessions on health (depression, self-esteem, anxiety, sleep, and pregnancy), relationships (kindness, generosity, relationships, change, appreciation, and acceptance) and performance (creativity, focus, happiness, and balance). The frequency and duration of usage will be in accordance to the instructions of the app.
  Arms: Headspace Application Treatment Group

SUMMARY:
The study is a prospective, randomized, non-blinded comparative group clinical trial comparing participants who receive access to a mindfulness software app, Headspace, to those who receive standard care (i.e., a list of resources on mindfulness and health). It is hypothesized that participants randomized to the Headspace mindfulness application will exhibit greater improvement in HbA1C and quality of life measures compared to those randomized to standard care.

DETAILED DESCRIPTION:
Stress has been associated with diabetes mellitus, and is believed to both precipitate the onset and disrupt the control of diabetes. The overall quality of life, measured as physical and social functioning and perceived as physical and mental well-being, has been shown to be adversely impacted in those living with diabetes compared to people with no chronic illness. Both the physiological effects of poorly managed diabetes and the psychological stress of dealing with chronic illness can have negative tolls on the physical, social and mental well-being of the patient.

Although the emotional problems in diabetic patients have received increasing attention in the recent decade, these issues often remain unrecognized in clinical practice and untreated. Previous research suggest that antidepressant medication and cognitive behavioral therapy can be effective in the treatment of major depression in a proportion of diabetic patients; however, the use of these medications is often accompanied by side effects, lack of response to medication, or relapse. One accessible group intervention that proved successful in reducing emotional distress and improving quality of life in nonpatients and patient groups is mindfulness-based cognitive therapy. The central component of such intervention is the cultivation of mindfulness.

Mindfulness, the mental state of awareness of internal and external experiences, has been used as a technique in numerous types of therapies. Previous studies suggested that increased levels of mindfulness through mindfulness-based cognitive therapy mediated the effects of inventions on depressed and angry mood and stress in diabetes outpatients. Practice of mindfulness, such as meditation, has indicated correlation with well-being and perceived health, and that dispositional mindfulness may buffer against the negative impact of perceived stress on psychological well-being. Furthermore, mindfulness may be associated with better glucose regulation in diabetics, as individuals with higher levels of mindfulness may have a lower likelihood of obesity and greater sense of control. Hence, the role of mindfulness in the management of diabetes warrants further investigations.

A promising digital health platform, Headspace, provides guided meditation sessions, mindfulness training, meditation resources via a software application. Headspace has already been used in a number of clinical trials exploring the effects of mindfulness training. For instance, one study examining the impact of mindfulness on workplace stress found significant increases in well-being and perceived job control, and reductions in anxiety, depressive symptoms, diastolic blood pressure and sleep problems.

The objective of this study is to determine the effectiveness of using the Headspace mindfulness application compared to the standard care of providing resources on mindfulness to patients with diabetes. Specifically, the study will test the hypothesis that participants randomized to the Headspace app group will exhibit greater improvement in HbA1C and quality of life measures compared to those randomized to standard care.

Participants randomized to mindfulness app group will be given 3 months of free access to Headspace, a digital service that provides guided meditation sessions and mindfulness training. Headspace consists of video sessions on the foundations of mindfulness, health, relationships and performance. Participants randomized to standard care will not receive Headspace, but instead, a list of resources on mindfulness and health, until the 3-month study is complete.

At the 3-month visit, participants in both groups will have HbA1C taken and quality of life questionnaire completed. No further data will be collected after the final 3-month visit. At this time, participants in the control group will receive the same 3-month access to Headspace as if the participants had been randomized to the treatment group, for equality purposes.

ELIGIBILITY:
Inclusion Criteria:

* Provides full informed consent to participate in the study
* Established diagnosis of diabetes mellitus according to Canadian Diabetes Association criteria at the time of screening for the study
* Has an age ≥12 years
* Has a most recent HbA1C measurement of ≥8%
* Has access to an electronic device that supports Headspace (i.e., tablet or smart phone)

Exclusion Criteria:

* Has a most recent HbA1C measurement of <8%
* Has a physical disability or psychiatric diagnosis which would limit the ability to adhere to the study regimen, as judged by the investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C | 3 months
  A hypothesized reduction in HbA1C by 3 months post-randomization in participants in the treatment group compared to control group.
Quality of life | 3 months
  A hypothesized improvement in quality of life measurements, assessed by SD36 questionnaire, by 3 months post-randomization in participants in the treatment group compared to control group.

SECONDARY OUTCOMES:
Medication adherence | 3 months
  Assessed with Diabetes Distress Screening Scale
Social support | 3 months
  Assessed with Diabetes Distress Screening Scale
Diabetes empowerment | 3 months
  Assessed with Diabetes Distress Screening Scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bradley C. Stress and diabetes. Handbook of Life Stress, Cognition and Health. New York: John Wiley & Sons 1988:383-401.
- [Background] Rubin RR, Peyrot M. Quality of life and diabetes. Diabetes Metab Res Rev. 1999 May-Jun;15(3):205-18. doi: 10.1002/(sici)1520-7560(199905/06)15:33.0.co;2-o. PMID 10441043
- [Background] Kan C, Silva N, Golden SH, Rajala U, Timonen M, Stahl D, Ismail K. A systematic review and meta-analysis of the association between depression and insulin resistance. Diabetes Care. 2013 Feb;36(2):480-9. doi: 10.2337/dc12-1442. PMID 23349152
- [Background] Tunceli K, Bradley CJ, Nerenz D, Williams LK, Pladevall M, Elston Lafata J. The impact of diabetes on employment and work productivity. Diabetes Care. 2005 Nov;28(11):2662-7. doi: 10.2337/diacare.28.11.2662. PMID 16249536
- [Background] Pouwer F, Beekman AT, Lubach C, Snoek FJ. Nurses' recognition and registration of depression, anxiety and diabetes-specific emotional problems in outpatients with diabetes mellitus. Patient Educ Couns. 2006 Feb;60(2):235-40. doi: 10.1016/j.pec.2005.01.009. PMID 16442465
- [Background] Pouwer F. Should we screen for emotional distress in type 2 diabetes mellitus? Nat Rev Endocrinol. 2009 Dec;5(12):665-71. doi: 10.1038/nrendo.2009.214. Epub 2009 Nov 3. PMID 19884900
- [Background] Segal ZV, Williams JMG, Teasdale JD. Mindfulness-Based Cognitive Therapy for Depression: A New Approach to Preventing Relapse. New York, Guilford Press, 2002.
- [Background] Haenen S, Nyklicek I, van Son J, Pop V, Pouwer F. Mindfulness facets as differential mediators of short and long-term effects of Mindfulness-Based Cognitive Therapy in diabetes outpatients: Findings from the DiaMind randomized trial. J Psychosom Res. 2016 Jun;85:44-50. doi: 10.1016/j.jpsychores.2016.04.006. Epub 2016 Apr 22. PMID 27212669
- [Background] van Son J, Nyklicek I, Pop VJ, Blonk MC, Erdtsieck RJ, Spooren PF, Toorians AW, Pouwer F. The effects of a mindfulness-based intervention on emotional distress, quality of life, and HbA(1c) in outpatients with diabetes (DiaMind): a randomized controlled trial. Diabetes Care. 2013 Apr;36(4):823-30. doi: 10.2337/dc12-1477. Epub 2012 Nov 27. PMID 23193218
- [Background] Branstrom R, Duncan LG, Moskowitz JT. The association between dispositional mindfulness, psychological well-being, and perceived health in a Swedish population-based sample. Br J Health Psychol. 2011 May;16(Pt 2):300-16. doi: 10.1348/135910710X501683. Epub 2011 Mar 8. PMID 21489058
- [Background] Loucks EB, Gilman SE, Britton WB, Gutman R, Eaton CB, Buka SL. Associations of Mindfulness with Glucose Regulation and Diabetes. Am J Health Behav. 2016 Mar;40(2):258-67. doi: 10.5993/AJHB.40.2.11. PMID 26931758
- See also: Current study examining the impact of mindfulness on workplace stress found significant increases in well-being and perceived job control, and reductions in anxiety, depressive symptoms, diastolic blood pressure and sleep problems. — https://clinicaltrials.gov/ct2/show/study/NCT01661569